CLINICAL TRIAL: NCT05414162
Title: Multiparametric Cardiac MRI in Oncological Patients Under Chimeric Antigen Receptor T-Cell Therapy
Brief Title: Multiparametric Cardiac MRI in Patients Under CAR T-cell Therapy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Bonn (Other)
Responsible Party: Principal Investigator, Julian Alexander Luetkens, Head of Cardiovascular Imaging, Principal Investigator, Senior Physician, University Hospital, Bonn
Other Study IDs: 81/22
Record Dates: First submitted 2022-06-07; First posted 2022-06-10 (Actual); Last update posted 2022-06-15 (Actual); Status verified 2022-06

CONDITIONS: DLBCL; Multiple Myeloma; Cytokine Release Syndrome; Myocarditis; CAR T-cell Therapy; ALL; PCBCL; Follicular Lymphoma; MCL
Keywords: Cardiac; MRI; CAR T-cell therapy; Myocarditis; CRS
MeSH Terms: conditions — Multiple Myeloma; Cytokine Release Syndrome; Myocarditis; Lymphoma, Follicular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No

GROUPS / COHORTS (1):
- CAR T-cell Therapy Group: Hematooncological patients undergoing CAR T-cell therapy with Tisagenlecleucel, Axicabtagen-ciloleucel, Idecabtagen-vicleucel, Brexucabtagene autoleucel, Lisocabtagene maraleucel or Ciltacabtagene Autoleucel (dosages, frequency and duration to be determined by the treating oncologist).
  Interventions: Diagnostic Test: Cardiac MRI

INTERVENTIONS:
Diagnostic Test: Cardiac MRI — Hematooncology patients under CAR T-cell therapy will receive 3 MRI examinations: at baseline, within 2 weeks of start of CAR T-cell therapy, and at 6 months follow-up.

SUMMARY:
Recently chimeric antigen receptor (CAR) T-cell therapy, a new class of chemo therapy, has gained regulatory approval for the treatment of diseases such as B-cell lymphoma. Known side effects include cytokine release syndrome, which has been described to lead to myocarditis, but larger studies exploring this relationship are currently lacking. In this prospective study, the investigators aim to explore the potential effects of CAR T-cell therapy using cardiac MRI on the heart.

DETAILED DESCRIPTION:
Genetically modified chimeric antigen receptor (CAR) T cells specifically targeting CD19 or "B cell maturation antigen" (BCMA) have shown remarkable advances in the treatment of highly refractory and relapsing hematological malignancies including diffuse large B-cell lymphoma or multiple myeloma. However, this potent therapy is hampered by serious, potentially life threatening complications, which might also involve the cardiovascular system. The potential cardiotoxic profile remains poorly defined and insufficiently understood. This proposal describes a prospective, longitudinal, intraindividual cardiac magnetic resonance imaging (MRI) study in oncological patients, which are scheduled for CAR T cell therapy for cancer treatment. This explorative study is designed to evaluate and monitor acute and late effects of CAR T cell therapy on the heart muscle. Systematic cardiac MRI monitoring correlated with the clinical course and thorough immunological assessment is the next step in helping to understand the extent, pattern, and pathophysiology of CAR T cell therapy related cardiovascular adverse events.

A chimeric antigen receptor (CAR) is a recombinant fusion protein that activates T cells upon recognition of a specific antigen on the cell surface of target cells. Therapeutic success was especially noticed with CD19-specific CAR T cells in the treatment of highly refractory and relapsing hematological malignancies. CD19 is an effective target due to its expression throughout the development line of B cells and has a frequent and high-level expression on the surface of nearly all B-cell malignancies. In addition, it is not found on other normal tissue cells, including the heart, and is not shed as a soluble form. The process of manufacturing CAR T cells typically requires 3 to 4 weeks. Autologous T cells are first collected from the patient and then genetically modified ex vivo with lentiviral or retroviral vectors to reprogram the T cells to recognize tumor cells expressing a tumor associated antigen (e.g., CD19 or BCMA). The CAR T cells a multiplied in large quantities before being administered to the patient within a single infusion. Before the infusion of CAR T cells, patients undergo lymphodepleting chemotherapy, most commonly with a combination of fludarabine and cyclophosphamide. This suppresses the patient's endogenous T cell compartment and allows an in vivo expansion of the transferred CAR T cells. Although the CAR T cell therapy has clearly advanced the treatment of highly refractory or relapsing hematological malignancies, there are potentially severe drawbacks of this therapy. One especially worrisome shortcoming is the potential therapy association with the unique toxicities of a cytokine release syndrome (CRS) and neurologic toxicities.

Cardiovascular complications associated with CAR T cell therapy are less well defined but can be subclassified into autoimmune toxicities resulting from antigen-specific T cell infiltration of the heart and cytokine-mediated toxicities. Cytokine-associated cardiotoxicities have been reported especially in the setting of CRS and might be the cause for most of the observed cardiovascular side effects. In a retrospective study from Alvi et al. cardiovascular events were systematically investigated in adults treated with CAR T cell therapy. The study included 137 patients and found that up to 12% of patients had clinical apparent cardiovascular events after CAR T cell therapy initiation (median time to event 21 days). Cardiovascular events included cardiovascular death, new onset heart failure, decompensated heart failure, and new onset of arrhythmia. A decrease in left ventricular function was observed in 28% of patients while 54% of patients had an elevated troponin. Interestingly, all cardiovascular events occurred in patients with grade ≥ 2 CRS and 95% of events occurred after troponin elevation. Another retrospective study from Lefebvre et al. investigated the occurrence of major adverse cardiovascular events (MACE) in 145 adult patients treated with CAR T cell therapy. MACE included cardiovascular death, symptomatic heart failure, acute coronary syndrome, ischemic stroke, and new onset arrhythmias. In total, 31 out of 145 (21%) patients had MACE at a median time of 11 days after CAR T cell infusion. MACE was independently associated with CRS grade 3 or 4 and baseline creatinine. Overall survival after one year was 71%. Another retrospective study analyzing 116 patients with serial echocardiograms after CAR T cell therapy found that 10% of patients developed a new cardiomyopathy with a decrease of left ventricular ejection fraction (average decrease from 58% to 37%), mostly observed in patients with grade ≥ 2 CRS. Another study with a patient pool of 126, found that 10% of patients developed severe cardiac disorders after CAR T cell therapy including new onset heart failure, acute coronary syndrome, and myocardial infarction.

Cardiac MRI for assessment of acute and chronic cardiac effects in CAR T cell therapy As the impact and the pathophysiology of cardiotoxicity of CAR T cell therapies to the heart is poorly understood, it is still unclear, whether cardiotoxicity is simply an early phenomenon associated with the cytokine storm within the scope of the CRS or whether there are more direct cardiotoxic effects from the CAR T cells themselves. It has also been proposed that the observed systolic dysfunction in this setting is a sequalae of a stress induced Takotsubo syndrome. In this context, the physiological stress from the CRS could trigger the occurrence of Takotsubo syndrome. To explore the extent of cardiac injury and inflammation and the pattern of myocardial involvement related to CAR T cell therapy, cardiac MRI must be considered as the imaging modality of choice, particularly due to its inherent capabilities of advanced tissue characterization. Cardiac MRI can characterize myocardial tissue alterations, analyze involvement patterns, and give important insights into the remodeling processes. To date, no cardiac MRI studies in patients with CAR T cell therapy exist. However, in this context, multiparametric cardiac MRI can be used to detect and quantify acute diffuse myocardial tissue alterations, such as myocardial edema and fibrosis. Furthermore, alterations in myocardial function can be detected with high sensitivity by using myocardial strain analysis. Late gadolinium enhancement imaging has a very high specificity for the detection of necrotic inflammatory lesions, especially in the context of inflammatory cardiomyopathies, and could directly show inflammatory lesions associated with CAR T cell therapy. Also, cardiac MRI could reliably identify different patterns of wall motion abnormalities which are associated with Takotsubo syndrome (i.e., apical, midventricular, basal or focal types). A recent study from our group in patients under immune checkpoint inhibitors (ICI) for cancer treatment suggests that cardiac MRI is able to show subtle therapy related treatment effects and can support evidence of a specific imaging pattern of ICI-related myocarditis. Also, cardiac MRI is the imaging modality of choice to show longterm, cardiotoxic effects of chemotherapy. It is considered the reference standard for measurement of ventricular volumes and function making it ideally suited to assess adverse cardiac remodeling after termination of cancer treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing CAR T-cell therapy
* Consent to participate in study

Exclusion Criteria:

* Inability to undergo MRI examinations due to large metallic implants, cardiac pacemakers/neurostimulators, or claustrophobia
* Known cardiac conditions such as status post heart attack or myocarditis, complex congenital heard disease, or cardiomyopathies.
* Birth control using an IUD.
* Pregnancy or breastfeeding.
* Renal insufficiency with a GFR below 30 ml/min/1.73m2

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with a histopathologically confirmed B-cell lymphoma or multiple myeloma who are planned for CAR T-cell therapy who fulfill the inclusion and exlcusion criteria will be recruited.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2022-05-16 (Actual); Primary Completion 2024-05 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Extent and pattern of acute cardiac effects of CAR T-cell therapy | 2 weeks
  To investigate to what extent and with which patterns CAR T cell therapy leads to acute cardiac effects in terms of inflammation, fibrosis, and myocardial dysfunction that can be detected with cardiac MRI.
Long-term cardiac remodeling effects of CAR T-cell therapy | 6 months
  To explore whether CAR T cell therapy leads to long-term cardiac remodeling effects in terms of inflammation, fibrosis, and myocardial dysfunction that can be detected with cardiac MRI.
Correlate MRI findings with clinical course | 6 months
  To assess whether changes in cardiac MRI parameters obtained from objectives 1 and 2 correlate with the clinical course (e.g., CRS development), cytokines and immunological markers and might predict major adverse cardiac events (MACE).

CONTACTS AND LOCATIONS:
Overall Officials: Julian Luetkens, MD, Principal Investigator — University Hospital, Bonn; Annkristin Heine, MD, Principal Investigator — University Hospital, Bonn; Tobias Holderried, MD, Principal Investigator — University Hospital, Bonn; Dmitrij Kravchenko, MD, Principal Investigator — University Hospital, Bonn
Locations (1):
- University Hospital Bonn, Bonn, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Gross G, Waks T, Eshhar Z. Expression of immunoglobulin-T-cell receptor chimeric molecules as functional receptors with antibody-type specificity. Proc Natl Acad Sci U S A. 1989 Dec;86(24):10024-8. doi: 10.1073/pnas.86.24.10024. PMID 2513569
- [Background] Razeghian E, Nasution MKM, Rahman HS, Gardanova ZR, Abdelbasset WK, Aravindhan S, Bokov DO, Suksatan W, Nakhaei P, Shariatzadeh S, Marofi F, Yazdanifar M, Shamlou S, Motavalli R, Khiavi FM. A deep insight into CRISPR/Cas9 application in CAR-T cell-based tumor immunotherapies. Stem Cell Res Ther. 2021 Jul 28;12(1):428. doi: 10.1186/s13287-021-02510-7. PMID 34321099
- [Background] Mohanty R, Chowdhury CR, Arega S, Sen P, Ganguly P, Ganguly N. CAR T cell therapy: A new era for cancer treatment (Review). Oncol Rep. 2019 Dec;42(6):2183-2195. doi: 10.3892/or.2019.7335. Epub 2019 Sep 24. PMID 31578576
- [Background] Sermer D, Brentjens R. CAR T-cell therapy: Full speed ahead. Hematol Oncol. 2019 Jun;37 Suppl 1:95-100. doi: 10.1002/hon.2591. PMID 31187533
- [Background] Yanez L, Alarcon A, Sanchez-Escamilla M, Perales MA. How I treat adverse effects of CAR-T cell therapy. ESMO Open. 2020 Aug;4(Suppl 4):e000746. doi: 10.1136/esmoopen-2020-000746. PMID 32839196
- [Background] Lee DW, Santomasso BD, Locke FL, Ghobadi A, Turtle CJ, Brudno JN, Maus MV, Park JH, Mead E, Pavletic S, Go WY, Eldjerou L, Gardner RA, Frey N, Curran KJ, Peggs K, Pasquini M, DiPersio JF, van den Brink MRM, Komanduri KV, Grupp SA, Neelapu SS. ASTCT Consensus Grading for Cytokine Release Syndrome and Neurologic Toxicity Associated with Immune Effector Cells. Biol Blood Marrow Transplant. 2019 Apr;25(4):625-638. doi: 10.1016/j.bbmt.2018.12.758. Epub 2018 Dec 25. PMID 30592986
- [Background] Afzal A, Farooque U, Gillies E, Hassell L. T-cell Therapy-Mediated Myocarditis Secondary to Cytokine Release Syndrome. Cureus. 2020 Aug 25;12(8):e10022. doi: 10.7759/cureus.10022. PMID 32983717
- [Background] Ganatra S, Redd R, Hayek SS, Parikh R, Azam T, Yanik GA, Spendley L, Nikiforow S, Jacobson C, Nohria A. Chimeric Antigen Receptor T-Cell Therapy-Associated Cardiomyopathy in Patients With Refractory or Relapsed Non-Hodgkin Lymphoma. Circulation. 2020 Oct 27;142(17):1687-1690. doi: 10.1161/CIRCULATIONAHA.120.048100. Epub 2020 Oct 26. No abstract available. PMID 33104402
- [Background] Ghosh AK, Chen DH, Guha A, Mackenzie S, Walker JM, Roddie C. CAR T Cell Therapy-Related Cardiovascular Outcomes and Management: Systemic Disease or Direct Cardiotoxicity? JACC CardioOncol. 2020 Mar 17;2(1):97-109. doi: 10.1016/j.jaccao.2020.02.011. eCollection 2020 Mar. PMID 34396213
- [Background] Luetkens JA, Doerner J, Thomas DK, Dabir D, Gieseke J, Sprinkart AM, Fimmers R, Stehning C, Homsi R, Schwab JO, Schild H, Naehle CP. Acute myocarditis: multiparametric cardiac MR imaging. Radiology. 2014 Nov;273(2):383-92. doi: 10.1148/radiol.14132540. Epub 2014 Jun 6. PMID 24910904
- [Background] Friedrich MG, Sechtem U, Schulz-Menger J, Holmvang G, Alakija P, Cooper LT, White JA, Abdel-Aty H, Gutberlet M, Prasad S, Aletras A, Laissy JP, Paterson I, Filipchuk NG, Kumar A, Pauschinger M, Liu P; International Consensus Group on Cardiovascular Magnetic Resonance in Myocarditis. Cardiovascular magnetic resonance in myocarditis: A JACC White Paper. J Am Coll Cardiol. 2009 Apr 28;53(17):1475-87. doi: 10.1016/j.jacc.2009.02.007. PMID 19389557
- [Background] Ferreira VM, Schulz-Menger J, Holmvang G, Kramer CM, Carbone I, Sechtem U, Kindermann I, Gutberlet M, Cooper LT, Liu P, Friedrich MG. Cardiovascular Magnetic Resonance in Nonischemic Myocardial Inflammation: Expert Recommendations. J Am Coll Cardiol. 2018 Dec 18;72(24):3158-3176. doi: 10.1016/j.jacc.2018.09.072. PMID 30545455
- [Background] Sprinkart AM, Luetkens JA, Traber F, Doerner J, Gieseke J, Schnackenburg B, Schmitz G, Thomas D, Homsi R, Block W, Schild H, Naehle CP. Gradient Spin Echo (GraSE) imaging for fast myocardial T2 mapping. J Cardiovasc Magn Reson. 2015 Feb 12;17(1):12. doi: 10.1186/s12968-015-0127-z. PMID 25885268
- [Background] Messroghli DR, Radjenovic A, Kozerke S, Higgins DM, Sivananthan MU, Ridgway JP. Modified Look-Locker inversion recovery (MOLLI) for high-resolution T1 mapping of the heart. Magn Reson Med. 2004 Jul;52(1):141-6. doi: 10.1002/mrm.20110. PMID 15236377
- [Background] Luetkens JA, Faron A, Isaak A, Dabir D, Kuetting D, Feisst A, Schmeel FC, Sprinkart AM, Thomas D. Comparison of Original and 2018 Lake Louise Criteria for Diagnosis of Acute Myocarditis: Results of a Validation Cohort. Radiol Cardiothorac Imaging. 2019 Jul 25;1(3):e190010. doi: 10.1148/ryct.2019190010. eCollection 2019 Aug. PMID 33778510
- [Background] Luetkens JA, Homsi R, Dabir D, Kuetting DL, Marx C, Doerner J, Schlesinger-Irsch U, Andrie R, Sprinkart AM, Schmeel FC, Stehning C, Fimmers R, Gieseke J, Naehle CP, Schild HH, Thomas DK. Comprehensive Cardiac Magnetic Resonance for Short-Term Follow-Up in Acute Myocarditis. J Am Heart Assoc. 2016 Jul 19;5(7):e003603. doi: 10.1161/JAHA.116.003603. PMID 27436306
- [Background] Kravchenko D, Isaak A, Zimmer S, Mesropyan N, Reinert M, Faron A, Pieper CC, Heine A, Velten M, Nattermann J, Kuetting D, Duerr GD, Attenberger UI, Luetkens JA. Cardiac MRI in Patients with Prolonged Cardiorespiratory Symptoms after Mild to Moderate COVID-19. Radiology. 2021 Dec;301(3):E419-E425. doi: 10.1148/radiol.2021211162. Epub 2021 Aug 10. PMID 34374593
- [Background] Luetkens JA, Doerner J, Schwarze-Zander C, Wasmuth JC, Boesecke C, Sprinkart AM, Schmeel FC, Homsi R, Gieseke J, Schild HH, Rockstroh JK, Naehle CP. Cardiac Magnetic Resonance Reveals Signs of Subclinical Myocardial Inflammation in Asymptomatic HIV-Infected Patients. Circ Cardiovasc Imaging. 2016 Mar;9(3):e004091. doi: 10.1161/CIRCIMAGING.115.004091. PMID 26951603
- [Background] Luetkens JA, von Landenberg C, Isaak A, Faron A, Kuetting D, Gliem C, Dabir D, Kornblum C, Thomas D. Comprehensive Cardiac Magnetic Resonance for Assessment of Cardiac Involvement in Myotonic Muscular Dystrophy Type 1 and 2 Without Known Cardiovascular Disease. Circ Cardiovasc Imaging. 2019 Jun;12(6):e009100. doi: 10.1161/CIRCIMAGING.119.009100. Epub 2019 May 29. No abstract available. PMID 31137956
- [Background] Gerhardt W, Ljungdahl L. Troponin T: a sensitive and specific diagnostic and prognostic marker of myocardial damage. Clin Chim Acta. 1998 Apr 6;272(1):47-57. doi: 10.1016/s0009-8981(97)00251-9. PMID 9581856
- [Background] Faron A, Isaak A, Mesropyan N, Reinert M, Schwab K, Sirokay J, Sprinkart AM, Bauernfeind FG, Dabir D, Pieper CC, Heine A, Kuetting D, Attenberger U, Landsberg J, Luetkens JA. Cardiac MRI Depicts Immune Checkpoint Inhibitor-induced Myocarditis: A Prospective Study. Radiology. 2021 Dec;301(3):602-609. doi: 10.1148/radiol.2021210814. Epub 2021 Sep 28. PMID 34581628
- [Background] Wang Y, Alkasab TK, Narin O, Nazarian RM, Kaewlai R, Kay J, Abujudeh HH. Incidence of nephrogenic systemic fibrosis after adoption of restrictive gadolinium-based contrast agent guidelines. Radiology. 2011 Jul;260(1):105-11. doi: 10.1148/radiol.11102340. Epub 2011 May 17. PMID 21586680
- [Background] Radbruch A, Weberling LD, Kieslich PJ, Hepp J, Kickingereder P, Wick W, Schlemmer HP, Bendszus M. High-Signal Intensity in the Dentate Nucleus and Globus Pallidus on Unenhanced T1-Weighted Images: Evaluation of the Macrocyclic Gadolinium-Based Contrast Agent Gadobutrol. Invest Radiol. 2015 Dec;50(12):805-10. doi: 10.1097/RLI.0000000000000227. PMID 26523910